CLINICAL TRIAL: NCT01814358
Title: Effects of Pre-meal Whey Protein Ingestion on Daily Glycemic Control and Oxidative Stress Mediated Postprandial Inflammation and Vascular Dysfunction Evoked by Consumption of a High-glycemic Meal
Brief Title: Whey Protein Effects on Gycemic Control and Vascular Function
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Thomas whey 01
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Blood Sugar (Glucose) Control; Blood Vessel (Vascular) Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Whey protein (Experimental): Subjects on this arm will receive whey protein
  Interventions: Dietary Supplement: Whey protein powder
- Gelatin protein (Active Comparator): Subjects on this arm will consume gelatin protein
  Interventions: Dietary Supplement: Control protein
- Control arm (No Intervention): Subjects on this arm will receive no intervention

INTERVENTIONS:
Dietary Supplement: Whey protein powder — Subjects on this arm will consume 20g whey protein powder mixed with water 15 minutes prior to breakfast, lunch, and dinner for two days
  Arms: Whey protein
Dietary Supplement: Control protein — Subjects on this arm will consume 20g gelatin protein powder mixed with water 15 minutes prior to breakfast, lunch, and dinner for two days
  Arms: Gelatin protein

SUMMARY:
Risk for heart and blood vessel diseases is increased when blood sugar rises. Blood vessel dysfunction is common to such diseases. Elevated blood sugar after eating promotes blood vessel dysfunction. Dietary factors other than carbohydrates influence rises and falls in blood sugar. Dietary protein is associated with improved blood sugar control. Whey protein effectively blunts the rise in blood sugar after consuming a carbohydrate rich drink/meal in normal weight and obese adults. This study will investigate the efficacy of drinking a whey protein beverage prior to eating for improved daily blood sugar control in normal weight and obese adults in the "real world." Also, the study will test this dietary approach to reduce blood vessel dysfunction associated with eating a meal that causes blood sugar to rise. 24 normal weight and 24 obese men and premenopausal women (18-50y) will participate. Subjects will wear a sensor to monitor daily blood sugar changes in response to their typically consumed diets for 2 days. Subjects will report to the UCLA CTRC the morning after the monitoring period for measurement of blood vessel function after eating a breakfast cereal meal. Blood samples will be obtained before and after the meal to measure relevant health markers. Subjects will repeat the 2-day diet and breakfast cereal meal challenge after a week or more, and will consume either a chocolate flavored 1) whey protein or 2) gelatin protein (control) shake prior to each meal. Neither subjects nor researchers will know which protein ("double blind"). Subjects will receive the alternate protein intervention after another week or more ("crossover"). We think drinking the protein shake prior to meals will reduce daily blood sugar rises and falls after eating and blunt the blood vessel dysfunction that results from eating the breakfast cereal.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* BMI between 18.5 and 25 or ≥ 30
* Willingness to provide written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding currently or in prior 6 months
* Menopause in women
* Regular consumption of > 1 serving per day of milk/yogurt
* Known heart arrhythmia
* Use of tobacco products
* Any disease/pathological condition known to influence outcomes
* Use of medications/dietary supplements known to influence outcomes
* Recent or planned changes in diet/exercise

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Average 24 hour glucose | 48 hours
  The 24-hour glucose level (average of 48-hour monitoring period) for whey protein arm compared to other protein arm

SECONDARY OUTCOMES:
Glycemic variability | 48 hours
Post-meal percent change Brachial Artery Flow Mediated Dilation (FMD) | 120 minutes
Post-meal monocyte inflammatory signaling | 60 minutes
Post-meal percent change femoral artery blood flow (FBF) | 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Thomas, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States